CLINICAL TRIAL: NCT02680912
Title: Warm Needle Acupuncture vs. Needle Acupuncture for Osteoarthritis of the Knee: A Pilot Study
Brief Title: Warm Needle Acupuncture vs Needle Acupuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London South Bank University (Other)
Collaborators: British Acupuncture Council (Other); Confucius Institute for Traditional Chinese Medicine, London South Bank University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6505
Record Dates: First submitted 2016-02-04; First posted 2016-02-12 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Bi syndrome
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Warm needle acupuncture (Experimental): Warm needle acupuncture (wenzhen; 温针) is where moxa cones are placed on the handle of the needle, after the needle has been inserted. Once lit, heat transmits along the shaft of the needle to the acupuncture point.
  Moxa refers to the herb mugwort (Artemisia vulgaris) that is burnt to warm specific parts of the body, including acupuncture points.
  Interventions: Device: Warm needle acupuncture
- Basic needle acupuncture (Active Comparator): Basic needle acupuncture is the use of acupuncture needles alone, without other methods of stimulation.
  Interventions: Device: Needle acupuncture

INTERVENTIONS:
Device: Warm needle acupuncture — There will be 4-6 points used per knee, therefore 8-12 needles per treatment. Two points will be used as the core treatment ST 35 dubi, Ex-LE 5 xiyan. Four other acu-points can also be used from the following: Ahshi painful points local to the knee (locus dolendi), ST 36 zusanli, GB 34 yanglingquan, Sp 9 yinlingquan, ST34 liangqiu, Sp 10 xuehai, GB 33 yangxiguan, LR 7 xiguan, LR 8 ququan, heding Ex-LE 2 In addition to the acupuncture needles the warm needle acupuncture group will receive moxibustion on up to 4 points. Smokeless moxa will be used.
  Arms: Warm needle acupuncture
Device: Needle acupuncture — The point selection protocol will be exactly the same as the experimental group
  Arms: Basic needle acupuncture

SUMMARY:
This is a two-armed randomised controlled pilot study that investigates the component efficacy of moxibustion for osteoarthritis of the knee. Participants will be randomised to receive either warm needle acupuncture or needle acupuncture. Participants and acupuncturists will be blinded to group allocation. The primary and secondary outcome measures are WOMAC and SF36 respectively. Qualitative interviews will be used to gather information on the patients' experiences and perceptions of the trial and the treatment provided.

It is hypothesised that warm needle acupuncture will lead to a greater reduction in clinical signs and symptoms than needle acupuncture.

DETAILED DESCRIPTION:
Acupuncture Treatment

All participants will receive acupuncture. Only points local to the knee will be used. There will be 4-6 points used per knee, therefore 8 -12 needles per treatment. A record will be kept of the points used at each treatment. Both knees will be treated even if only one knee is painful. This will ensure that participants receive similar treatments.

Patients will be treated seated, as this allows better access to the relevant acupuncture points. It also helps ensure the moxibustion is carried out safely.

Participants will receive 8 treatments in the first 4 weeks (twice a week), then 4 treatments in 4 weeks (once a week).

Blinding procedures

The only difference in the procedures will be that lit cones are placed on the needles of the treatment group whilst unlit moxa cones will be placed on the needles of the control group. Smokeless moxa will be used. All patients will see the needles being inserted and the moxa cones placed on the needles by the acupuncturist. Skin guards will be placed at the base of the needle to reduce the immediate sense of heat on the surface of the skin. Similar skin guards are routinely used in acupuncture treatment to prevent any discomfort.

The acupuncturist will carry out a consultation at each session as per normal practice. After the needles have been inserted and the moxa cones have been placed on needles the acupuncturist leaves and an assistant acupuncturist enters the room. The assistant acupuncturist will place a screen in front of the patient to prevent them from seeing their knees. The assistant acupuncturist will then remove one cone at a time and light it. In the treatment group the lit cone is placed on the needle. In the control group the lit cone is place in a small dish close to the knee, a replacement unlit cone is placed on the needle. This process is repeated until all the cones are lit. The unlit cone is replaced on the needle of the control group to try and ensure they experience the same sensations as the treatment group. The use of a second acupuncturist to light the moxa ensures that the acupuncturist who carries out the consultation and inserts the needles is blinded to group allocation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain in at least one knee joint during the last six months.
* At baseline the WOMAC pain score must be ≥ 3 points (on a scale of 0-10)

In addition to the knee pain at least 3 of the following 6 must be present:

* Age > 50 years
* Stiffness < 30 minutes
* Crepitus
* Bony Tenderness
* Bony enlargement
* No palpable warmth

(ACR 2013)

Plus

* Ability to speak English
* Signed consent form

Exclusion Criteria:

* A systemic disease of the musculoskeletal system.
* Bone tumour, bone tumour like lesions or metastasis.
* Bone fracture in the lower extremities during the last three months.
* Acute infection or osteonecrosis in the knee joint.
* Recent sprain injury to the knee joint.
* Surgery of the afflicted extremity during the last six months or planned surgery.
* Ongoing cortico-steroid therapy or cortisone injections in the past six weeks.
* Taking anti-coagulant medication.
* Coagulopathy.
* Other pain condition that compels the patient to take analgesics for more than three days during the last four weeks.
* Addiction to analgesics, opiate or other drugs.
* Acupuncture treatment in the past 3 months.
* Dermatological disease within the acupuncture area impairing acupuncture treatment.
* Pregnant or breast-feeding patients.
* Inability to follow instructions or understand the consent form (insufficient command of language, dementia).
* Participation in another clinical study.
* Ongoing legal proceedings concerning degree of disability.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02; Primary Completion 2017-05-16 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Change from Baseline to follow up at 16 weeks

SECONDARY OUTCOMES:
SF36 (Rand) | Change from Baseline to follow up at 16 weeks
  Health Related Quality of Life (HRQL)

CONTACTS AND LOCATIONS:
Overall Officials: Ian K Appleyard, Principal Investigator — London South Bank University
Locations (1):
- Confucius Institute for TCM LSBU, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: WOMAC Osteoarthritis Index — http://www.womac.org/
- See also: ACR 2013, "Classification Criteria for Rheumatic Diseases: Idiopathic OA of the knee", American College of Rheumatology, [Online], , pp. 5 January 2014. — http://www.rheumatology.org/practice/clinical/classification/oaknee.asp